CLINICAL TRIAL: NCT00012467
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging, Phase II Study of the Safety and Antifungal Activity of Subcutaneous Recombinant Interferon-Gamma 1b (rIFN-Gamma 1b) in Conjunction With Standard Therapy in Patients With Acute Cryptococcal Meningitis
Brief Title: Safety and Antifungal Activity of Recombinant Interferon-Gamma 1b (rIFN-Gamma 1b) Given With Standard Therapy in Patients With Cryptococcal Meningitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: InterMune (Industry)
Responsible Party: Steven Porter, MD, PhD, InterMune Pharmaceuticals Inc.
Masking: Double | Purpose: Treatment
Other Study IDs: B013; GIMY-001
Record Dates: First submitted 2001-03-09; First posted 2001-08-31 (Estimated); Last update posted 2009-06-03 (Estimated); Status verified 2009-05

CONDITIONS: Meningitis, Cryptococcal; HIV Infections
Keywords: Interferon-gamma, Recombinant; Injections, Subcutaneous; Itraconazole; Dose-Response Relationship, Drug; Fluconazole; Flucytosine; Antifungal Agents; Amphotericin B; Meningitis, Cryptococcal
MeSH Terms: conditions — Meningitis, Cryptococcal; HIV Infections | interventions — Itraconazole; Flucytosine; Fluconazole; Amphotericin B; interferon gamma-1b

INTERVENTIONS:
Drug: Itraconazole
Drug: Flucytosine
Drug: Fluconazole
Drug: Amphotericin B
Drug: Interferon gamma-1b

SUMMARY:
The purpose of this study is to examine the antifungal activity of recombinant interferon-gamma 1b (rIFN-gamma 1b) given with standard antifungal therapy.

DETAILED DESCRIPTION:
Patients are randomized into 1 of 3 parallel groups for a 3-arm, 2-stage, double-blind and dose-ranging study for 14 weeks. In Stage 1, patients are hospitalized for 14 days of acute therapy. Patients receive rIFN-gamma 1b or placebo sc 3 times per week, intravenous (IV) AMB daily, and with or without oral 5-FC every 6 hours. Patients who have the ability to take oral medications, who do not have any significant clinical deterioration during the previous 14 days, and who meet the eligibility criteria can progress to Stage 2. In Stage 2 patients receive 84 days of consolidation therapy (56 days with study drug and 28 days of follow-up). On an outpatient basis, patients receive either placebo or 1 of 2 doses of rIFN-gamma 1b sc 3 times per week, and oral fluconazole daily or oral itraconazole 2 times a day.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for Stage 1 if they:

* Are at least 13 years old.
* Have consent of a parent, family member, or guardian if less than 18 years of age.
* Have cryptococcal meningitis for the first time or have had a relapse.
* Are not on any medications that cannot be taken with fluconazole or itraconazole, if the patient has trouble taking fluconazole.
* Patients may be eligible for Stage 2 if they:
* Had no serious decline in health, as determined by their doctor, during the previous 14 days (including mental health).
* Have received at least 7.5 mg/kg AMB in Stage 1.
* Have a positive CSF culture for C. neoformans.
* Can take oral medications.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Are in a coma.
* Are pregnant or breast-feeding.
* Are not using effective birth control methods, if able to have children.
* Are allergic to imidazole or triazole.
* Are allergic to rIFN-gamma 1b.
* Require drugs that are toxic to the kidneys, other than AMB.
* Received erythropoietin or red blood cell transfusions within 4 weeks of entering the study.
* Are receiving systemic corticosteroid therapy within 30 days of study or will require it during the study.
* Have had serious heart disease.
* Have had multiple sclerosis, peripheral vascular disease, or rheumatologic disorders.
* Have had disorders of the central nervous system (CNS) (not including emotional problems) or a seizure disorder, or have a current CNS disorder that would interfere with the study.
* Are receiving investigational therapy for C. neoformans within 90 days of starting the study drug.
* Have had more than 3 doses of AMB or more than 1200 mg of fluconazole or itraconazole as prior treatment and have begun current treatment for more than 72 hours prior to starting study medication. Fluconazole or itraconazole of no more than 200 mg daily is allowed.
* Are receiving AMB for C. neoformans within 30 days of starting treatment for the present episode.
* Are receiving rIFN-gamma 1b treatment within 90 days prior to starting the study drug.
* Have had therapy which affects the immune system within 30 days prior to starting the study drug.
* Are receiving investigational therapy for all other signs within 30 days prior to starting the study drug.
* Are not able to meet the study requirements, in the opinion of the investigator.
* Require chronic treatment with H2-blockers, and are able to receive only itraconazole in Stage 2.
* Show signs of or get treatment for another serious opportunistic infection within 4 weeks of starting the study drug.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2000-01; Study Completion 2001-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (7):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Washington Univ, St Louis, Missouri
  - UMDNJ - New Jersey Med School / Cooper Hosp, Camden, New Jersey
  - Univ of Med & Dentistry of New Jersey, Newark, New Jersey
  - Houston Veterans Administration Med Ctr, Houston, Texas
  - Univ of Texas / Med School at Houston, Houston, Texas
  - Audie L Murphy Veterans Administration Hosp, San Antonio, Texas
- Peru (2):
  - Hosp Nacional dos de Mayo, Lima
  - Instituto de Medicina Tropical, Lima